CLINICAL TRIAL: NCT05891626
Title: Group Intervention to Improve Vaccine Confidence and Vaccination in a Community Healthcare System: A Mixed Methods Study Design
Brief Title: Group Intervention on Vaccine Confidence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MultiCare Health System Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022/05/26
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Vaccination Refusal
Keywords: Vaccine confidence; Adult patient; Caregiver of pediatric patients; Missed opportunities for vaccination (MoV); Vaccination rates; Vaccine hesitancy
MeSH Terms: conditions — Vaccination Refusal; Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: cluster randomized controlled trial, mixed methods
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group intervention (Experimental): Six comparable general clinics (2 for pediatric care and 4 for adult primary care) from all MultiCare facilities will be selected to participate in the study. Half of the clinics will be in the Puget Sound Region and others in the Eastern Washington Areas. Allocation to the intervention will be based on randomization: one pediatric and two adult (Internal Medicine or Family Medicine) clinics will get the comprehensive intervention.
  Interventions: Behavioral: Group intervention
- Standard care (No Intervention): The other three facilities will stay as the control under routine care. The three control group sites will have no additional interventional activities regarding vaccination, except for MultiCare's usual vaccine promotion practices (which the interventional clinics will have also).

INTERVENTIONS:
Behavioral: Group intervention — An enhanced electronic reminder mechanism specialized on vaccines and actively highlight vaccine standing orders in the system.
  Set up a data benchmarks, so clinic managers or providers are able to aggregate immunization data, red flag missed opportunities, and facilitate modifying vaccine promotion plans.
  Other components:
  1. missed opportunities and doubts/hesitancy about immunization as a whole;
  2. specific questions with regard to specific vaccines;
  3. health conditions and socioeconomic/demographic vulnerabilities (insufficient resources in health literacy, linguistic or cultural considerations); and
  4. challenges in patient-clinician interactions. These components will be addressed through team training/meetings, pamphlets, physician-led speech in online videos, and group messages via MyChart on the clinic level.
  Arms: Group intervention

SUMMARY:
This study has one primary objective and two secondary objectives, with an overall goal of understanding barriers to vaccination and vaccination confidence, so that effective interventional strategies can be further developed and tested to improve vaccination outcomes in a community healthcare setting.

DETAILED DESCRIPTION:
The study will use a mixed methods approach, combining focus group discussion, virtual interviews with healthcare professionals, cross-sectional survey on vaccination attitude, and clinic-based intervention with a cluster randomized controlled trial design for the quantitative stage. They study will also follow up patients with interviews after the quantitative stage completes.

ELIGIBILITY:
Qualitative study standards:

Inclusion Criteria:

* having used MultiCare's services in the past 12 months or whose minor child(ren) has/have used MultiCare's services in the past 12 months, and who have been involved in the child(ren)'s immunization decision-making as a caregiver
* current residential location in Washington State
* willing to participate

Exclusion Criteria:

* terminal disease (to be decided)
* cognitive impairment
* main immune deficiency conditions

Quantitative study standards:

We will randomly (and) equally select clinics from 1) Puget Sound and 2) Eastern Washington areas. Since the intervention is on facility level (group intervention), instead of at patient level, blinding will also be impractical. We plan to use stratified random allocation within the pediatric (n1 = 2) or adult stratum (n2 = 4), to decide which sites will get the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 429 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Vaccine confidence scale(s) | 6 months over vaccination attitude for each subpopulation
  Vaccination attitude (confidence or hesitancy) measured by the following:
  For caregivers of 19-35 months children: Parent Attitudes about Childhood Vaccines Survey - Short Form (PACV-SF) and Emory Vaccine Confidence Index (EVCI);
  For caregivers of pediatric patients 3 years or older: Vaccination Confidence Scale (VCS) and EVCI;
  For adult patients: Vaccination Attitudes Examination Scale (VAX);
  For clinical workers/health professionals: VAX.

SECONDARY OUTCOMES:
Missed opportunities for vaccination (MOVs) | 6 months over vaccination attitude for each subpopulation
  Well visit completion in the previous 12 months prior to baseline, and post-pre changes in adult patients;
  Well-child visit completion rate 12 months prior to baseline, and post-pre changes in 3-18 yo for the pediatric clinics;
  Total numbers of well clinic visits at baseline and changes over 6 months.
Vaccination rates | 6 months over vaccination attitude for each subpopulation

CONTACTS AND LOCATIONS:
Locations (1):
- Jin, Puyallup, Washington, United States

IPD SHARING:
Plan to Share IPD: No